CLINICAL TRIAL: NCT02090361
Title: Efficacy of Collagen-elastin Dermal Substitute in the Treatment of Loss of Cutaneous Substances With Skin Grafts
Acronym: MATRIGREFFE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/008/HP
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Skin Graft; Collagen -Elastin Matrix
Keywords: collagen -elastin matrix; skin graft; loss of cutaneous substance
MeSH Terms: interventions — Skin Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- skin graft with dermal matrix (Experimental): Epidermization of the defect by applying a thin layer of autologous epidermis with addition of a dermal matrix
  Interventions: Procedure: skin graft
- skin graft - classic procedure (Placebo Comparator): Epidermization of the defect by applying a thin layer of autologous epidermis
  Interventions: Procedure: skin graft

INTERVENTIONS:
Procedure: skin graft — Epidermization of the defect by applying a thin layer of autologous epidermis

SUMMARY:
In reconstructive surgery , most losses of cutaneous substance require the use of a thin skin graft . This technique allows epidermization of the defect by applying a thin layer of autologous epidermis. It does not reconstitute the injured skin. Transplants cause retractile scars, adherent to the deep plan, that may require revision surgery . Since a decade , dermal matrices are mainly used in burned skin centers . The collagen -elastin matrix has the advantage to set up in the same operation that the skin graft and contain elastic fibers , two assets which improve the results of skin grafting.

Objective:

Evaluation of the clinical efficacy of the addition of a dermal matrix to skin graft on Skin Foldability, at day 360.

Methodology:

This is a multicenter randomized study (CHU Caen , Amiens, Rouen and Lille)

Conduct of the study :

The transplant will be performed according to the protocol defined between inter -region surgeons. The implementation of the dermal matrix will be in the same surgical technique as thin skin graft ( group 1 ) or the thin skin graft will be performed alone ( group 2) time .

Evaluation Criteria Main : Skin Foldability ( Uf ) assessed grafted site will be compared to the opposite side ungrafted evaluated at Day 360 . Quantitative data will be measured by a cutometer Skin Elasticity Meter 580 (Courage and Khazaba Electronic GmbH).

To achieve the main objective, it is planned to compare the ratio between Uf graft site and the opposite healthy site between two groups: skin + matrix graft , or skin graft only. Thus, the Wilcoxon test for independent samples will be used to settle bilateral formulation between the null hypothesis ( there is no difference between the two groups ) and the alternative hypothesis ( there is a difference between the two groups ) . In determining the overall risk of first species to 5% and the power of this test to detect the 90% expected under the alternative hypothesis difference should be the main criterion for evaluating at least 59 patients in each group so 118 patients total.

Prospect If the contribution of a dermal matrix in loss of skin substances improves skin pliability and reduces pain , functional and aesthetic sequelae grafts thin skin , the dermal matrix may be proposed as a complementary treatment in these indications.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Signed informed consent
* Patients with loss of cutaneous substance of at least 15 cm2
* Patient Without bone exposure, vascular, joint or tendon
* Eligibility for surgical treatment by skin graft
* Loss of substance trauma (avulsion, burns) or surgery (skin excision)

Exclusion Criteria:

* Patient with a chronic wound
* Wound superinfected
* Patient unable for local or general skin graft
* Patient with an old or a recent skin injury strictly contralateral to the graft site.
* Patient unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2014-06-18 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Skin Foldability ( Uf ) | Day 360
  Skin Foldability ( Uf ) will be assessed on grafted site compared to the opposite side ungrafted at day D360 . Quantitative data will be measured by a cutometer Skin Elasticity Meter 580 (Courage and Khazaba Electronic GmbH).

SECONDARY OUTCOMES:
Skin Foldability ( Uf ) | Day 180
  Skin Foldability ( Uf ) will be assessed on grafted site compared to the opposite side ungrafted at day D180 . Quantitative data will be measured by a cutometer Skin Elasticity Meter 580 (Courage and Khazaba Electronic GmbH)
Skin Foldability ( Uf ) | Day 90
  Skin Foldability ( Uf ) will be assessed on grafted site compared to the opposite side ungrafted at day D90 . Quantitative data will be measured by a cutometer Skin Elasticity Meter 580 (Courage and Khazaba Electronic GmbH)
Pain on the grafted site | D7
  Assessment of pain on the grafted site EVA at Day 7
pain on the grafted site | Day 15
  Assessment of pain on the grafted site at Day 15
pain on the grafted site | Day 30
  Assessment of pain at the grafted site EVA to D30
pain on the grafted site | Day 90
  Assessment of pain at the grafted site EVA at D30
pain on the grafted site | Day 180
  Assessment of pain at the grafted site EVA at Day 180
pain on the grafted site | Day 360
  Assessment of pain at the grafted site EVA at Day 360
tolerance of matriderm use | Day 360
  Occurrence within 360 days of a local complication requiring reoperation
Area healed | Day 7
  Evaluation of the percentage of area healed at Day 7
Area healed | Day 15
  Evaluation of the percentage of area healed at Day 15
Area healed | Day 30
  Evaluation of the percentage of area healed at Day 30
Assessment of functional effects | Day 30
  Assessment of functional effects of the scar on the patient 's daily activities defined at Day 30
Assessment of functional effects | Day 90
  Assessment of functional effects of the scar on the patient 's daily activities defined at Day 90
Assessment of functional effects | Day 180
  Assessment of functional effects of the scar on the patient 's daily activities defined at Day 180
Assessment of functional effects | Day 360
  Assessment of functional effects of the scar on the patient 's daily activities defined at Day 360
Aesthetic sequelae evaluation | Day 90
  Evaluation aesthetic sequelae by a committee of independent experts to study the photographs taken at day 90
Aesthetic sequelae evaluation | Day 180
  Evaluation aesthetic sequelae by a committee of independent experts to study the photographs taken at day 180
Aesthetic sequelae evaluation | Day 360
  Evaluation aesthetic sequelae by a committee of independent experts to study the photographs taken at day 360

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle AUQUIT-AUCKBUR, Pr, Principal Investigator — UH Rouen
Locations (4):
- France (4):
  - CHU d'Amiens, Amiens
  - CHU de Caen, Caen
  - CHU de Lille, Lille
  - UH Rouen, Rouen